CLINICAL TRIAL: NCT05229094
Title: EVA Nexus Field Observation Study. A Monocentric, Academic Field Observation Study of a Prototype of a New CE-labeled Vitrectomy Device Developed by DORC BV (The Netherlands).
Brief Title: EVA Nexus Vitrectomy Device Field Observation Study
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: 64913
Record Dates: First submitted 2021-12-24; First posted 2022-02-08 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Retina Disorder; Vitreous Disorder
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Eva Nexus — Eva Nexus vitrectomy device

SUMMARY:
determine the safety and effectiveness of the device.

DETAILED DESCRIPTION:
To perform a field observation study using the newly developed EVA Nexus vitrectomy device.

Patients that are scheduled for intra-ocular surgery regardless of the indication:

* Vitrectomy surgery
* Cataract surgery
* Vitrectomy combined with cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients that are scheduled for intra-ocular surgery regardless of the indication:
* Vitrectomy surgery
* Cataract surgery
* Vitrectomy combined with cataract surgery
* In case of (combined) vitrectomy: primary or repeat vitrectomy
* General or retrobulbar anesthesia, the latter can be combined with sedation
* Patients aged ≥ 18 years

Exclusion Criteria:

* Patients aged < 18 years

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients that are scheduled for intra-ocular surgery regardless of the indication:
  * Vitrectomy surgery
  * Cataract surgery
  * Vitrectomy combined with cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
to evaluate the intra-operative safety of a new surgical device | 2 days
  specific adverse events that may occur during the (phaco) vitrectomy will be recorded to assess the surgical safety.

SECONDARY OUTCOMES:
To evaluate the possible reduction of total surgical time | 1 day
  The time that was required to prepare the EVA Nexus will be recorded (connecting of supplies + priming).
To evaluate the impact of usage of the EVA NEXUS on the surgical parameters used during the procedure | 2 days
  The surgical parameters include a range of data collected on the following:
  Aspiration Irrigation / Infusion BSS Usage Vitrectomy Ultrasound Illumination Diathermy Micro-injection Silicone oil injection / extraction Laser
To evaluate possible (S)AE that may be related to the use of the surgical platform. | 2 days
  Rarely, adverse events (AE) that are related to the surgery may only become visible the day after the surgery. A postoperative check of the eye at the day after the surgery will be performed to determine the presence of such AE's.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, Phd, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peter S. Clinical trial to test the safety of the EVA Nexus surgical platform. Int J Retina Vitreous. 2024 Jun 24;10(1):45. doi: 10.1186/s40942-024-00563-3. PMID 38915097

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT05229094/Prot_SAP_000.pdf